CLINICAL TRIAL: NCT04179331
Title: Neurotensin Infusions in Healthy Individuals - Effects on Appetite, Food Intake, Hormone Secretions and Cardiovascular Responses
Brief Title: Neurotensin Infusions in Healthy Individuals -
Acronym: NIHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Simon Veedfald, Primary investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NT-2-19
Record Dates: First submitted 2019-11-07; First posted 2019-11-27 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Appetite regulation; Food intake; Ad libitum; Hormone secretion
MeSH Terms: interventions — Neurotensin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Acute physiological experiments conducted in healthy individuals in a University Hospital setting.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded. Neither the investigators performing the experiments or the participants know the nature of the intervention on the two study days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurotensin (Experimental)
  Interventions: Other: Neurotensin
- Saline (Experimental)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Neurotensin — Neurotensin is an endogenous peptide released from the distal small intestine. It will be administered at three doses (2.5, 5.0 and 7.5pmol/kg/min), each for 1h, in sequence.
  Arms: Neurotensin
Other: Saline — Isotonic saline will serve as a placebo.
  Arms: Saline

SUMMARY:
Neurotensin (NT) is a gut peptide released postprandially from the small intestine. It is known to exert a range of enterogastrone effects and in animal models it reduces food intake when administered by parenteral routes.

In this study, after a 1h baseline period, three doses (2.5, 5.0 and 7.5pmol/kg/min) of NT will be administered in sequence each infusion lasting 1h. On a placebo day saline will be infused similarly 1h infusions. During the final infusion (7.5pmol/kg/min) an ad libitum meal will be ingested. During the experiments blood samples will be collected and subjective perceptions recorded using validated visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* Age = or above 18 years
* normal haemoglobin levels
* male
* Informed consent

Exclusion Criteria:

* Diabetes mellitus (fasting plasma glucose or HbA1c)
* Familiy history of diabetes mellitus
* Intestinal disease (incl e.g. inflammatory bowel disease and malabsorbtion)
* Family history of inflammatory bowel disease
* Previous intestinal resection
* Body mass index (BMI) over 25 kg/m2
* Smoker
* Nephropathy (S-creatinine> 130 μM)
* Liver disease (ALAT and/or ASAT > 2 × upper normal limit)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Food intake | From time point t=190-220 minutes
  The amount of food ingested over 30 minutes will be determined.

SECONDARY OUTCOMES:
Hunger | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Satiation | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Fullness | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Prospective food intake | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Comfort | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Thirst | -45, -15, 15, 45, 75, 105, 135, 165, 220, 250 minutes
  Visual analogue scale (100mm)
Neurotensin | -60, -30, -15, 0, 15, 30, 60, 75, 90, 120, 135, 150, 180, 220 minutes
  plasma concentration (intact and total)
Pancreatic polypeptide | -60, -30, -15, 0, 15, 30, 60, 75, 90, 120, 135, 150, 180, 220 minutes
  Plasma concentration (intact and total)
Glucagon | -60, -30, -15, 0, 15, 30, 60, 75, 90, 120, 135, 150, 180, 220 minutes
  Plasma concentration
insulin and C-peptide | -60, -30, -15, 0, 15, 30, 60, 75, 90, 120, 135, 150, 180, 220 minutes
  Serum concentration
Heart rate | -60 to 250 minutes
  Pulse rate every 10 min
Blood pressure | -60 to 250 minutes
  Systolic and diastolic blood pressures (mmHg) every 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- hvidovre Hospital, Hvidovre, Capital, Denmark